CLINICAL TRIAL: NCT03200899
Title: Computer Assisted Cognitive Rehabilitation for Persons With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Alexa Stuifbergen, Professor and Dean, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2008-10-0101
Record Dates: First submitted 2017-06-21; First posted 2017-06-27 (Actual); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Multiple Sclerosis
Keywords: cognitive rehabilitation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Care providers are not informed of the participant's participation in a particular arm. Staff collecting outcome data are not aware of the participant's assignment to intervention or usual care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Memory, Attention, Problem Solving Skills in MS (MAPSS-MS) (Experimental): Participants randomized to this arm receive the MAPSS-MS intervention. The MAPSS-MS is an an 8 week computer assisted cognitive rehabilitation intervention. The group based component of the intervention emphasizes use of compensatory cognitive strategies as well as lifestyle modifications to enhance cognition. Participants also complete home computer training (minimum 3 times per week for 45 minutes) using a special suite of games designed by Lumosity.
  Interventions: Behavioral: MAPSS-MS
- Usual Care plus Computer games (Active Comparator): Participants randomized to this arm receive usual care and are referred to MY BRAIN GAMES web site.
  Interventions: Other: Usual Care plus computer games

INTERVENTIONS:
Behavioral: MAPSS-MS — MAPSS-MS is a computer-assisted cognitive rehabilitation intervention. It is a combination of home computer training and 8-weeks of group sessions on lifestyle change and compensatory cognitive strategies.
  Arms: Memory, Attention, Problem Solving Skills in MS (MAPSS-MS)
Other: Usual Care plus computer games — Participants assigned to this arm receive their usual medical care and referral to the "My Brain Games" website.
  Arms: Usual Care plus Computer games

SUMMARY:
The effects of multiple sclerosis (MS) on cognition, thought to occur in 50-75% of persons with MS, have gained increasing recognition as one of the major disabling symptoms of the disease. While numerous studies have addressed the emotional and physical impact of MS, little attention has been given to strategies that might help manage the cognitive changes commonly experienced by persons with MS. The proposed study will test a novel computer-assisted cognitive rehabilitation intervention, MAPSS-MS (Memory, Attention, & Problem Solving Skills for Persons with MS). The MAPSS-MS integrates the powerful effects of group interventions to build self-efficacy for new cognitive compensatory strategies/behaviors with individual home-based computer-assisted training. The computer training will assist individuals to develop cognitive skills that they can apply to everyday life using the compensatory strategies learned in the class sessions. In the recently completed exploratory study with 61 persons with MS (R21NR011076), the eight-week MAPSS-MS intervention was acceptable and feasible and had medium to large effects on the use of compensatory strategies and performance on neuropsychological tests of verbal memory. The proposed study will test the refined MAPSS-MS intervention with a larger more diverse sample (N=180) across multiple sites, extend the period of post-intervention follow-up to 6 months and establish whether performance improvements on neuropsychological tests make the important transfer to improved neuro-cognitive functioning in everyday life.

The specific aims of this study are to: (1) Evaluate the efficacy of the novel MAPSS-MS cognitive rehabilitation intervention to improve overall neuro-cognitive competence in activities of daily living including verbal memory performance, use of compensatory cognitive strategies and performance on cognitive-related instrumental activities of daily living (IADL) among persons with MS; (2) Evaluate the efficacy of the MAPSS-MS intervention to improve self-efficacy and related aspects of cognitive performance (non-verbal learning/memory, information processing speed and attention, verbal fluency and complex scanning and tracking) among persons with MS; and (3) Determine the number of intervention participants who achieve and maintain their self-identified cognitive goals three and six months following the intervention. The effects of the intervention on outcome variables will be assessed using a randomized controlled trial design with a comparison group receiving usual care computer games. Measurements of study variables will occur at baseline, immediately after the MAPSS-MS intervention, and three months and six months after the intervention is complete. Statistical analysis will include descriptive statistics and HLM analysis to account for the nested design. The intent-to-treat approach will be used.

Public Health Statement: This research will provide new knowledge about an innovative intervention to improve memory, use of compensatory strategies, and performance of cognitive activities and instrumental activities of daily living for persons with MS. If effective, the intervention would provide a new and feasible approach to target a serious, debilitating problem commonly experienced by persons with MS.

ELIGIBILITY:
Inclusion Criteria:

* Clinically definite diagnosis of MS;
* Age 18 to 60;
* Capable of understanding and complying with the study protocol;
* Able to read and write in English;
* Visual acuity of at least 20/70 with correction in order to work on the computer screen;
* Stable disease at the time of entry into the study (relapse free for at least 90 days);
* Subjective concerns about their cognitive functioning (based on the Perceived Deficits Questionnaire); and
* Home internet access;

Exclusion Criteria:

* Other medical causes of dementia or other neurological disorders that may impact cognition or emotions;
* Evidence of major psychiatric disorder; or
* Major functional limitations that preclude them from participating in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 183 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexa Stuifbergen, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data files will be de-identified and data will be available on request to the investigators - estimated availability 2020
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: WIll be shared on request in 2020 and beyond
Access Criteria: Qualified investigators with IRB approval

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from three large metropolitan communities in Texas: Houston, San Antonio and Dallas. Participants were recruited via physician referral, targeted mailings to persons with MS on the mailing list of the National MS Society, contact with support groups, and notices in MS newletters and websites.
Period: Overall Study
Arm/Group | Memory, Attention, Problem Solving Skills in MS (MAPSS-MS) | Usual Care Plus Computer Games
Started | 93 | 90
T2 - Immediately Post-intervention | 85 | 78
T3 - 3-months Post-intervention | 82 | 74
Completed | 83 | 67
Not Completed | 10 | 23
Not completed — Lost to Follow-up | 10 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Memory, Attention, Problem Solving Skills in MS (MAPSS-MS) | Usual Care Plus Computer Games | Total
Number analyzed (Participants) | 93 | 90 | 183
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 93 | 90 | 183
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (7.5) | 49.4 (8.5) | 49.6 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 80 | 160
  Male | 13 | 10 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 9 | 18
  Not Hispanic or Latino | 84 | 81 | 165
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 17 | 34
  White | 73 | 64 | 137
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 3 | 8 | 11
Region of Enrollment [Number; unit: participants]
  United States | 93 | 90 | 183
Marital Status [Count of Participants; unit: Participants]
  Married | 56 | 61 | 117
  Un-married | 37 | 29 | 66
Employment Status [Count of Participants; unit: Participants]
  Full-time | 25 | 28 | 53
  Part-time | 5 | 3 | 8
  Unemployed - Disability | 32 | 39 | 71
  Retired | 12 | 5 | 17
  Other | 8 | 2 | 10
  Not reported | 11 | 13 | 24
Years Since Diagnosis [Mean (Standard Deviation); unit: years] | 13.9 (8.05) | 12.1 (8.07) | 13.0 (8.08)
MS Type [Count of Participants; unit: Participants]
  Benign Sensory | 3 | 3 | 6
  Relapsing-Remitting | 64 | 61 | 125
  Primary Progressive | 3 | 5 | 8
  Secondary Progressive | 14 | 10 | 24
  Progressive-Relapsing | 1 | 1 | 2
  Unable to choose one/don't know | 8 | 9 | 17
  Not reported | 0 | 1 | 1
Expanded Disability Status Scale (EDSS) [Mean (Standard Deviation); unit: units on a scale] — Expanded Disability Status Scale. This is an ordinal scale with scores ranging from 0 to 9.5. Higher scores indicate greater functional impairment.
  units on a scale | 5.1 (1.63) | 5.3 (1.5) | 5.2 (1.56)

OUTCOME MEASURES:

1. Primary Outcome: Neuro-cognitive Competence in Daily Living - California Verbal Learning Test-II
Description: Verbal memory performance (verbal learning and remembering) as measured by performance on the California Verbal Learning Test II (CVLT-II). Total score represents the number of words recalled from a 16 item list over 5 trials. Higher scores represent greater verbal learning and remembering. Scores can range from 0 to 80.
Time Frame: 6 months post-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memory, Attention, Problem Solving Skills in MS (MAPSS-MS) | Usual Care Plus Computer Games
Number analyzed (Participants) | 93 | 90
units on a scale | 56.1 (12.9) | 53.6 (12.9)
Statistical Analysis 1: Comparison: Memory, Attention, Problem Solving Skills in MS (MAPSS-MS) vs Usual Care Plus Computer Games; Test type: Superiority; p = 0.926, ANCOVA

2. Primary Outcome: Use of Compensatory Cognitive Strategies
Description: Scores on the Strategy Subscale of the Multi-Factorial Memory Memory Questionnaire. The subscale includes 19 various memory aids and strategies and respondents are asked to rate how frequently they used each strategy during the past 2 weeks using a 5 point scale (never to all the time). Scores can range from 0 to 76. HIgher scores indicate greater use of compensatory memory strategies.
Time Frame: 6 months post-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memory, Attention, Problem Solving Skills in MS (MAPSS-MS) | Usual Care Plus Computer Games
Number analyzed (Participants) | 93 | 90
units on a scale | 40.2 (11.0) | 39.5 (11.2)
Statistical Analysis 1: Comparison: Memory, Attention, Problem Solving Skills in MS (MAPSS-MS) vs Usual Care Plus Computer Games; Test type: Superiority; p = 0.750, ANCOVA

3. Primary Outcome: Cognitive-related Instrumental Activities of Daily Living (IADL) Among Persons With MS
Description: Scores on the Everyday Problems Test - Revised (EPT-R). This scale assess the cognitive ability to reason and solve problems encountered in daily living. The revised version included 30 items and scores can range from 0 to 30. HIgher scores indicate better performance on problem solving.
Time Frame: 6 months post intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memory, Attention, Problem Solving Skills in MS (MAPSS-MS) | Usual Care Plus Computer Games
Number analyzed (Participants) | 93 | 90
units on a scale | 24.2 (4.8) | 23.5 (4.4)
Statistical Analysis 1: Comparison: Memory, Attention, Problem Solving Skills in MS (MAPSS-MS) vs Usual Care Plus Computer Games; Test type: Superiority; p = 0.129, ANCOVA

4. Secondary Outcome: Self-Efficacy
Description: Scores on the 17 item general self-efficacy scale. Respondents rate their confidence in their ability to affect outcomes in various contexts and situations using a 5-point Likert scale. Scores can range from 17 to 85 with higher scores representing greater perceived self-efficacy expectations.
Time Frame: 6 months post intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memory, Attention, Problem Solving Skills in MS (MAPSS-MS) | Usual Care Plus Computer Games
Number analyzed (Participants) | 93 | 90
units on a scale | 63.7 (11.1) | 61.1 (12.0)
Statistical Analysis 1: Comparison: Memory, Attention, Problem Solving Skills in MS (MAPSS-MS) vs Usual Care Plus Computer Games; Test type: Superiority; p = 0.152, ANCOVA

5. Secondary Outcome: Verbal Fluency
Description: Controlled Oral Word Association Test (COWAT) is a measure of verbal fluency and word finding. It requires participants to generate words from initial letters (normally F, A and S) under time constraints, normally 60 seconds per letter. The score reflects the number of words generated across the trials and can vary from 0 to the maximum number generated. Higher scores reflect a greater number of words and greater fluency and word finding.
Time Frame: 6 months post intervention
Measure: Mean (Standard Deviation); unit: words generated
Arm/Group | Memory, Attention, Problem Solving Skills in MS (MAPSS-MS) | Usual Care Plus Computer Games
Number analyzed (Participants) | 93 | 90
words generated | 39.5 (12.1) | 36.9 (11.9)
Statistical Analysis 1: Comparison: Memory, Attention, Problem Solving Skills in MS (MAPSS-MS) vs Usual Care Plus Computer Games; Test type: Superiority; p = 0.037, ANCOVA

6. Secondary Outcome: Nonverbal Learning and Memory
Description: Brief Visuospatial Memory Test, 2nd ed (BVMT-R) asses visuospatial memory and was used as a measure of non-verbal learning and memory. The total recall score was used in this study and this score represents the sum of all valid items generated across learning trials 1-3.
  In each trial, 0-12 points can be obtained. The recognition (yes/no) is scored by one or zero points with a maximum of 12 points. The total score for the total recall ranges from 0 to 36. HIgher scores indicate better memory and recall.
Time Frame: 6 months post intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memory, Attention, Problem Solving Skills in MS (MAPSS-MS) | Usual Care Plus Computer Games
Number analyzed (Participants) | 93 | 90
units on a scale | 21.9 (7.0) | 20.1 (6.7)
Statistical Analysis 1: Comparison: Memory, Attention, Problem Solving Skills in MS (MAPSS-MS) vs Usual Care Plus Computer Games; Test type: Superiority; p = 0.297, ANCOVA

7. Secondary Outcome: Auditory Information Processing Speed and Flexibility
Description: The Paced Auditory Serial Addition Test (PASAT) - 3 second was used as the measure of auditory information processing speed and flexibility. Scores represent the number of correct responses during the 3 minute test and can range from 0 to 60. Higher scores indicate better information processing speed and flexibility.
Time Frame: 6 months post intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memory, Attention, Problem Solving Skills in MS (MAPSS-MS) | Usual Care Plus Computer Games
Number analyzed (Participants) | 93 | 90
units on a scale | 47.6 (11.9) | 45.9 (11.8)
Statistical Analysis 1: Comparison: Memory, Attention, Problem Solving Skills in MS (MAPSS-MS) vs Usual Care Plus Computer Games; Test type: Superiority; p = 0.293, ANCOVA

8. Secondary Outcome: Psychomotor Processing Speed
Description: The Symbol Digit Modalities Test (SDMT) was used to measure psychomotor processing speed, complex scanning and visual tracking. Respondents have 90 seconds to pair digits/numbers with abstract geometric symbols. Total scores represent the number of correct matches within the time period and can range from 0 to 110. Higher scores reflect better information processing speed.
Time Frame: 6 months post intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memory, Attention, Problem Solving Skills in MS (MAPSS-MS) | Usual Care Plus Computer Games
Number analyzed (Participants) | 93 | 90
units on a scale | 54.6 (12.2) | 52.0 (12.4)
Statistical Analysis 1: Comparison: Memory, Attention, Problem Solving Skills in MS (MAPSS-MS) vs Usual Care Plus Computer Games; Test type: Superiority; p = 0.045, ANCOVA

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Memory, Attention, Problem Solving Skills in MS (MAPSS-MS) | Usual Care Plus Computer Games
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/90
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/90
Other Adverse Events (participants affected / at risk) | 0/93 | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-07): https://cdn.clinicaltrials.gov/large-docs/99/NCT03200899/Prot_SAP_000.pdf